CLINICAL TRIAL: NCT01366664
Title: A Randomized, Double-blind, Placebo-Controlled, Crossover Study Assessing the Pharmacodynamic Effects of Dapoxetine Concomitantly Administered in Subjects Taking Terazosin
Brief Title: A Pharmacodynamic Study of Dapoxetine Concomitantly Administered in Participants Taking Terazosin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR018607; R096769PRE1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Ejaculation
Keywords: Premature Ejaculation; Selective Serotonin Reuptake Inhibitor; Dapoxetine; PRILIGY; Terazosin; Pharmacodynamic; Pharmacokinetic
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Treatment sequence 1 Treatment Period 1 (stable dose of terazosin [2 to 10 mg] + dapoxetine 60 mg administered orally once daily for 5 days) followed up to 14 days later by Treatment Period 2 (stable dose of terazosin [2 to 10 mg] + placebo administered orally once daily for 5 days)
  Interventions: Drug: Treatment sequence 1
- 002 (Experimental): Treatment sequence 2 Treatment Period 1 (stable dose of terazosin [2 to 10 mg] + placebo administered orally once daily for 5 days) followed up to 14 days later by Treatment Period 2 (stable dose of terazosin [2 to 10 mg] + dapoxetine 60 mg administered orally once daily for 5 days)
  Interventions: Drug: Treatment sequence 2

INTERVENTIONS:
Drug: Treatment sequence 2 — Treatment Period 1 (stable dose of terazosin [2, 5, or 10 mg] + placebo administered orally once daily for 5 days) followed up to 14 days later by Treatment Period 2 (stable dose of terazosin [2, 5, or 10 mg] + dapoxetine 60 mg administered orally once daily for 5 days)
  Arms: 002
Drug: Treatment sequence 1 — Treatment Period 1 (stable dose of terazosin [2, 5, or 10 mg] + dapoxetine 60 mg administered orally once daily for 5 days) followed up to 14 days later by Treatment Period 2 (stable dose of terazosin [2, 5, or 10 mg] + placebo administered orally once daily for 5 days)
  Arms: 001

SUMMARY:
The purpose of this study is to assess the pharmacodynamics (the actions or effects a drug has on the body), pharmacokinetics (blood levels), safety, and tolerability of dapoxetine 60 mg when concomitantly administered in participants taking terazosin.

DETAILED DESCRIPTION:
This is a multiple-center, randomized (participants are assigned to study drug by chance), multiple-dose, double-blind (neither physician nor participant knows the treatment assigned), placebo (inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled, 2-period crossover (participants may receive different interventions sequentially during the trial) study to assess the pharmacodynamics, pharmacokinetics, safety, and tolerability of dapoxetine when concomitantly administered in adult male participants who have been on a stable dose of terazosin or doxazosin for at least 6 weeks. Study drugs used will be terazosin (a drug given for the treatment of hypertension and benign prostatic hyperplasia) and dapoxetine (a new drug being studied for the treatment of premature ejaculation). This study consists of a screening phase followed by a double-blind, placebo-controlled treatment phase consisting of 2 treatment periods. Participants will remain on their prescribed dose of terazosin and participants taking doxazosin will be converted to terazosin using the protocol-defined dose conversion (including assessment of control of urinary symptoms and risk for urinary retention). Participants will be administered concomitant (at the same time) dapoxetine or placebo once daily. Blood samples for pharmacodynamic and pharmacokinetic measurements will be collected at selected times during the study. Safety will be monitored. The total duration of study participation will be approximately 49 days. Participants will remain on their prescribed dose of terazosin (2 to 10 mg taken once daily by mouth) and will be administered daily by mouth concomitant dapoxetine 60 mg or placebo doses during 2 treatment periods (each 7 days in duration conducted in the study center). A period of up to 14 days will separate the treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* On a stable regimen of terazosin (2 to 10 mg) or doxazosin (2 to 8 mg) taken daily for at least 6 weeks for the treatment of hypertension or benign prostatic hyperplasia
* a body mass index between 18 and 35 kg/m², inclusive
* a body weight of not less than 50 kg
* supine (laying down) blood pressure measurements between 90 and 150 mmHg, inclusive
* and, diastolic blood pressure measurements no higher than 95 mmHg.

Exclusion Criteria:

* History of current clinically significant illness or any other illness that the investigator considers should exclude the study participant or that could interfere with the interpretation of study results
* symptomatic orthostatic hypotension (a decrease of >=20 mm Hg systolic blood pressure measured after 2 but before 3 minutes after changing from supine (laying down) to standing position)
* taking a medication that is known to cause orthostatic hypotension, other than terazosin
* and, taking more than 2 other antihypertensive medications or taking an antihypertensive medication that is excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference between standing and supine blood pressure measurements | Days 1-2
Difference between standing and supine blood pressure measurements | Days 5-6

SECONDARY OUTCOMES:
Plasma concentrations of dapoxetine | Blood samples collected prior to and for 24 hours following dapoxetine/placebo administration on Days 1 and 5 of each treatment period and prior to dosing on Days 3 and 4
Plasma concentrations of dapoxetine metabolite desmethyldapoxetine | Blood samples collected prior to and for 24 hours following dapoxetine/placebo administration on Days 1 and 5 of each treatment period and prior to dosing on Days 3 and 4
Number and type of adverse events | Up to a Maximum of 26 Days
Clinical laboratory test values | Up to a Maximum of 26 Days
Physical examination findings | Up to a Maximum of 26 Days
Vital sign measurements | Up to a Maximum of 26 Days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- United States (6):
  - Anniston, Alabama
  - Tempe, Arizona
  - Costa Mesa, California
  - Miramar, Florida
  - Knoxville, Tennessee
  - Dallas, Texas

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study Assessing the Pharmacodynamic Effects of Dapoxetine Concomitantly Administered in Subjects Taking Terazosin — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1119&filename=CR018607_CSR.pdf